CLINICAL TRIAL: NCT06606613
Title: Midurethral Sling Versus Cross-linked Hyaluronic Acid/dextranomer (CLHA/Dx) for the Treatment of Stress Urinary Incontinence
Brief Title: Cross-linked Hyaluronic Acid/dextranomer for the Treatment of Stress Urinary Incontinence
Acronym: (CLHA/Dx)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, İBRAHİM KARACA, Associate Proffesor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170924
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Urinary Stress Incontinence (SI)
Keywords: Cross-linked hyaluronic acid/dextranomer; Mid-urethral sling; Female; Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective before-after (pre-post) interventional study, in which the effectiveness and safety of intraurethral cross-linked hyaluronic acid/dextranomer injection in female stress urinary incontinence patients were compared with those undergoing mid-urethral sling procedures.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraurethral injection group (Experimental): Intraurethral Cross-linked hyaluronic acid/dextranomer injection was performed in female patients with Stress Urinary incontinence
  Interventions: Procedure: Intraurethral injection
- Mid-urethral sling group (Active Comparator): Mid-urethral sling procedure was performed in female patients with Stress Urinary incontinence
  Interventions: Procedure: Mid-urethral sling

INTERVENTIONS:
Procedure: Intraurethral injection — Procedure: Intraurethral injection
  Patients are positioned in the lithotomy position during the procedure. General and/or local anesthesia is administered depending on the investigator's preference. An applicator developed for intraurethral injection will be used. This device comprises a holder that is placed into and fixates the urethra (i.e., it distends the urethral circumference, thus smoothing out the longitudinal folds), allowing the use of four syringes to inject cross-linked hyaluronic acid/dextranomer at approximately the 2, 4, 8, and 10 o'clock positions.
  Drug: Cross-linked hyaluronic acid/dextranomer
  Arms: Intraurethral injection group
Procedure: Mid-urethral sling — Procedure: Starting with the dorsal lithotomy position, a foley catheter is inserted to the urethra. Starting with 1-1.5 cm below the urethral meatus, a 1.5-2 cm vertical incision is made. Following the dissection of anterior vaginal mucosa, pubocervical fascia should be dissected sharply .
  Dissection is continued laterally to the ischiopubic ramus. Starting downwards from the tendinous insertion of the adductor longus muscle at the level of clitoris, a 1cm incision is made close to the bone. The needle is placed in to the incision and passed medially through the obturator membrane. It has to be considered that the needle is passed very close to the bone in order not to damage the obturator vessel-nerve bundle. With the guidance of the opposite hand's index finger in the vaginal incision the tip of the needle has to be palpated afterwards passing with a 45-degree angle rotation. The next manoeuvre is passing the tip of the needle beside the urethra through the vaginal incision .
  Arms: Mid-urethral sling group

SUMMARY:
The investigators aimed to evaluate the effectiveness and safety of intraurethral cross-linked hyaluronic acid/dextranomer (CLHA/Dx) injection for the treatment of stress urinary incontinence (SUI) in women.

DETAILED DESCRIPTION:
This single-center prospective pre-post interventional study was conducted between October 2025 and April 2025 with 60 women . Quality of life was evaluated with the Incontinence Quality of Life Scale (I-QoL) and the lower urinary tract symptoms of women were evaluated with the International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS). Incontinence status was assessed via the Stamey Incontinence Grade scale. The need for additional treatment (re-injection, other surgical approaches, etc.) was recorded.

Participants were followed up to 6 months after intervention. All outcomes of interest and complications were evaluated/recorded at three preplanned visits (postoperative 1st, 3rd, 6th, months).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stress Urinary Incontinence.
* Presence of incontinence during the Valsalva maneuver.
* Positive Marshall-Marchetti test result.
* Post-void residual urine volume of ≤100 mL.

Exclusion Criteria:

* Temporary urinary incontinence.
* Delirium.
* Urinary tract infection.
* Urethritis.
* Pure urge incontinence.
* Nocturnal enuresis.
* Decreased bladder compliance or detrusor contraction observed in urodynamic -studies.
* Leakage of urine with low bladder pressure.
* Psychiatric conditions (severe depression and anxiety).
* Body mass index (BMI) > 35 kg/m².
* Use of medications that may influence bladder storage or emptying.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Need for addtional treatment within the 3st month | Within the 3 st month
  Patients who are needed to treat with re-injection or other surgical approaches.
Need for addtional treatment within the 1st month | Within the 1st month
  Patients who are needed to treat with re-injection or other surgical approaches
Need for addtional treatment within the 6 st month | Within the 6 st month
  Patients who are needed to treat with re-injection or other surgical approaches
Presence of complication within 6 months after intervention | Within 6 months after intervention
  Presence of complication such as infection at injection site, urinary tract infection, hematuria, persistent pain, de novo urge incontinence) in all patients.
Change in the Stamey Incontinence Grade at 6months | Change from baseline at 6months.
  All patients were evaluated as follows: Grade 0: No incontinence; Grade 1: Incontinence with coughing or straining; Grade 2: Incontinence with change in position or walking; Grade 3: Total incontinence at all times.Stamey grading is specifically a 4-level scale of incontinence severity, ranging from 0 (continent/dry) to 3 (total incontinence, regardless of activity)
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 3 | Change from baseline at 3 month
  All patients were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.The ICIQ-FLUTS consists of 12 questions related to LUTS divided into three areas: filling (4 questions), voiding (3 questions), and incontinence (5 questions). The answers are based on experiences with LUTS in the previous four weeks. The score is calculated by domain and it ranges from zero to ten in each question. As the score increases, the severity of the symptom increases.
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 1 month | Change from baseline at 1 month
  All patients were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.The ICIQ-FLUTS consists of 12 questions related to LUTS divided into three areas: filling (4 questions), voiding (3 questions), and incontinence (5 questions). The answers are based on experiences with LUTS in the previous four weeks. The score is calculated by domain and it ranges from zero to ten in each question. As the score increases, the severity of the symptom increases.
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 6 month | Change from baseline at 6 month
  All patients were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.The ICIQ-FLUTS consists of 12 questions related to LUTS divided into three areas: filling (4 questions), voiding (3 questions), and incontinence (5 questions). The answers are based on experiences with LUTS in the previous four weeks. The score is calculated by domain and it ranges from zero to ten in each question. As the score increases, the severity of the symptom increases.
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 3 months | Change from baseline at 3 month
  All patients were evaluated İth. the I-QOL which has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).The I-QOL is divided into 3 subscales:Avoidance and limiting behavior (ALB),Psychosocial impact (PSI),Social embarrassment (SE). Subjects use a 5-point response scale with values ranging from 1 (extremely) to 5 (not at all). A mean score for each subscale is calculated (averaging the scores for the items in each subscale) as well as a total score for all 22 items (sum of all subscale scores).The scores are then transformed to a 'Scale score' ranging from 0-100 points for ease of interpretation: Scale score = (sum of the items - lowest possible score)/possible raw score range X 100.
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 6 months | Change from baseline at 6 month
  All patients were evaluated with the I-QOL which has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).The I-QOL is divided into 3 subscales:Avoidance and limiting behavior (ALB),Psychosocial impact (PSI),Social embarrassment (SE). Subjects use a 5-point response scale with values ranging from 1 (extremely) to 5 (not at all). A mean score for each subscale is calculated (averaging the scores for the items in each subscale) as well as a total score for all 22 items (sum of all subscale scores).The scores are then transformed to a 'Scale score' ranging from 0-100 points for ease of interpretation: Scale score = (sum of the items - lowest possible score)/possible raw score range X 100.
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 1 month | Change from baseline at 1 month
  All patients were evaluated with the I-QOL which has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).The I-QOL is divided into 3 subscales:Avoidance and limiting behavior (ALB),Psychosocial impact (PSI),Social embarrassment (SE). Subjects use a 5-point response scale with values ranging from 1 (extremely) to 5 (not at all). A mean score for each subscale is calculated (averaging the scores for the items in each subscale) as well as a total score for all 22 items (sum of all subscale scores).The scores are then transformed to a 'Scale score' ranging from 0-100 points for ease of interpretation: Scale score = (sum of the items - lowest possible score)/possible raw score range X 100.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Bakircay University, Izmir, BAYRAKLI, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol